CLINICAL TRIAL: NCT01602822
Title: A Phase IV Open-label Evaluation of Safety, Tolerability and Patient Acceptance of Atazanavir Boosted With Ritonavir Combined With a Fixed-dose Formulation of Tenofovir DF and Emtricitabine for nPEP Following Potential Exposure to HIV-1
Brief Title: Safety and Acceptability Study of Non-occupational Prophylaxis (PEP) Following Potential Exposure to HIV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Grade 3 elevation in liver function tests
Sponsor: Kenneth H. Mayer, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry); Gilead Sciences (Industry); Abbott (Industry)
Responsible Party: Sponsor-Investigator, Kenneth H. Mayer, MD, Medical Director, The Fenway Institute, Fenway Community Health
Organization: Fenway Community Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BMS PEP
Record Dates: First submitted 2012-02-08; First posted 2012-05-21 (Estimated); Results first posted 2025-04-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: HIV
Keywords: HIV Prevention; Non-occupational Post-Exposure Prophylaxis (NPEP); Post-Exposure Prophylaxis (PEP)
MeSH Terms: interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Open-label phase IV study of a new regimen for antiretroviral post-exposure prophylaxis
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atazanavir, Ritonavir, Truvada (Other): Tenofovir DF and Emtricitabine; Ritonavir-boosted Atazanavir
  Interventions: Drug: Tenofovir DF and Emtricitabine; Ritonavir-boosted Atazanavir

INTERVENTIONS:
Drug: Tenofovir DF and Emtricitabine; Ritonavir-boosted Atazanavir — TDF 300mg and FTC 200mg fixed-dose combination tablet (TDF/FTC) once daily, and atazanavir, one 300mg tablet and one 100 mg ritonavir given once daily
  Other Names: Truvada

SUMMARY:
This study will evaluate how safe and tolerable a combination of taking three-drugs will be for the purpose of preventing HIV transmission after a high-risk sexual contact exposure in HIV uninfected adults.

DETAILED DESCRIPTION:
Participants are given a regimen containing tenofovir disoproxil fumarate (TDF) 300mg and emtricitabine (FTC) 200mg fixed-dose combination tablet (TDF/FTC) once daily, and atazanavir, one 300mg tablet and one 100 mg ritonavir given once daily,for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 at time of first visit.
2. HIV uninfected on the basis of a negative HIV Rapid Test
3. Possible non-occupational exposure to HIV-1, recent enough to permit receiving the first dose of study medication within 72 hours from the end of the exposure.

Exclusion Criteria:

1. Women who are actively trying to become pregnant.
2. Pregnancy and/or Breastfeeding.
3. Known self report of Chronic Hepatitis B infection or prior antiretroviral therapy for hepatitis B.
4. Known intolerance or allergy to study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Mayer, MD, Principal Investigator — Fenway Health
Locations (1):
- Fenway Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
De-identified participant data describing the adverse events will be available for review upon request

REFERENCES:
- See also: Fenway Health homepage — http://www.fenwayhealth.org/site/PageServer

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atazanavir, Ritonavir, Truvada
Started | 11
Completed | 0
Not Completed | 11
Not completed — Adverse Event | 11

BASELINE CHARACTERISTICS:
Population: Men and women who present within 72 hours of a potential non-occupational exposure to HIV-1.
Arm/Group | Atazanavir, Ritonavir, Truvada
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 37 [23 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Safety of Regimen - Symptoms
Description: Number of subjects who experienced moderate-to-severe symptoms on the symptom-directed physical exam at or before visit 3.
Time Frame: Visit 3- Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Atazanavir, Ritonavir, Truvada
Number analyzed (Participants) | 11
Participants
  None or Mild | 4
  Moderate to Severe | 7

2. Primary Outcome: Safety of Regimen - Adverse Events/Serious Adverse Events Considered Related
Description: Number of subjects who experience adverse or serious adverse events that are considered related to the use of the drug regimen at or before visit 3.
Time Frame: visit 3 - day 30
Measure: Number; unit: participants
Arm/Group | Atazanavir, Ritonavir, Truvada
Number analyzed (Participants) | 11
participants
  No related events | 4
  1 or more related adverse/serious advers events | 7

3. Primary Outcome: Safety of Regimen - Unsafe Biological Test
Description: Number of subjects who have an unsafe biological test result as part of the laboratory screen for safety levels (e.g., CBC, Creatinine, etc.) at or before visit 3.
Time Frame: visit 3 - day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Atazanavir, Ritonavir, Truvada
Number analyzed (Participants) | 11
Participants
  no unsafe lab tests | 4
  1 or more unsafe lab tests | 7

4. Secondary Outcome: Awareness of NPEP
Description: Assess awareness as measured by how many participants had initially heard of NPEP prior to the incident exposure
Time Frame: Visit 2- Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Atazanavir, Ritonavir, Truvada
Number analyzed (Participants) | 11
Participants
  number of participants who had heard of nPEP prior to exposure | 10
  Number of participants who had not heard of nPEP prior to exposure | 1

5. Secondary Outcome: Adherence Rate - Overall
Description: Adherence to the regimen will be assessed by whether the regimen was completed as prescribed or not. χ2 tests will be used to assess differences in the proportion of both completion and adherence between participants in the current study and participants in previous studies of NPEP at Fenway Health (historical controls).
Time Frame: Visit 3- Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Atazanavir, Ritonavir, Truvada
Number analyzed (Participants) | 11
Participants
  Non-Adherent (30 day) | 7
  Adherent (30 day) | 4

6. Secondary Outcome: Prior nPEP Use
Description: Number of participants who had used nPEP prior to participation in the study.
Time Frame: Visit 2- Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Atazanavir, Ritonavir, Truvada
Number analyzed (Participants) | 11
Participants
  Number of participants who had used nPEP in their lifetime prior to participating in this study | 2
  Number of participants who had not used nPEP in their lifetime prior to participating in this study. | 9

7. Secondary Outcome: Adherence - Degree of Adherence
Description: Number of participants who completed prescribed regimen
Time Frame: Visit 1- Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Atazanavir, Ritonavir, Truvada
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Arm/Group | Atazanavir, Ritonavir, Truvada
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 7/11
Other Adverse Events (participants affected / at risk) | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atazanavir, Ritonavir, Truvada (N=11)
Grade 3 elevation in liver function tests (Hepatobiliary disorders) | 7 (11) — Due to the Grade 3 and Grade 4 elevations in liver function tests, the study was terminated on 22 May 2012
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atazanavir, Ritonavir, Truvada (N=11)
jaundice (Gastrointestinal disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Study terminated early as a result of Grade 3 and Grade 4 elevations in liver function tests

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No